CLINICAL TRIAL: NCT01350128
Title: A Randomized, Double-Blind, Chronic Dosing (7 Days), Three-Period, Six-Treatment, Placebo-Controlled, Incomplete Block, Cross-Over, Multi-Center Study to Assess Efficacy and Safety of Four Doses of PT001 in Patients With Moderate to Severe COPD, Compared With Atrovent® HFA Inhalation Aerosol (Open-Label) as An Active Control
Brief Title: PT001 MDI Versus Atrovent Study in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT001002
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PT001 MDI (Dose 1) (Experimental): PT001 MDI
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 2) (Experimental): PT001 MDI
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 3) (Experimental): PT001 MDI
  Interventions: Drug: PT001 MDI
- PT001 MDI (Dose 4) (Experimental): PT001 MDI
  Interventions: Drug: PT001 MDI
- Ipratropium Bromide HFA Inhalation Aerosol (Active Comparator): Ipratropium Bromide HFA Inhalation Aerosol
  Interventions: Drug: Ipratropium Bromide HFA Inhalation Aerosol
- Placebo MDI (Placebo Comparator): PT001 Placebo MDI
  Interventions: Other: Placebo MDI

INTERVENTIONS:
Drug: PT001 MDI — PT001 MDI administered as two puffs BID for 7 days
  Arms: PT001 MDI (Dose 1); PT001 MDI (Dose 2); PT001 MDI (Dose 3); PT001 MDI (Dose 4)
Drug: Ipratropium Bromide HFA Inhalation Aerosol — Taken as 2 inhalations of the 17 µg per actuation strength MDI QID
  Other Names: Atrovent
  Arms: Ipratropium Bromide HFA Inhalation Aerosol
Other: Placebo MDI — Matching placebo to PT001 MDI administered as two puffs BID for 7 days
  Arms: Placebo MDI

SUMMARY:
The overall objective of this study is to determine an optimal dose and dosing regimen of PT001 MDI for further evaluation in later stage studies.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate efficacy relative to placebo of PT001 MDI in patients with moderate to severe chronic obstructive pulmonary disease (COPD) within the range of doses evaluated in this protocol. To this end, each dose of PT001 MDI will be compared to placebo with respect to the primary efficacy endpoint, FEV1 AUC0-12 relative to baseline.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Clinical history of COPD with airflow limitation that is not fully reversible
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post- bronchodilator FEV1/FVC ratio of < or = 0.70
* A measured post- bronchodilator FEV1 > or = 750ml or 30% predicted and < or = 80% of predicted normal values
* Able to change COPD treatment as required by protocol

Key Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 3 months of Screening
* Clinically significant medical conditions that preclude participation in the study (e.g. clinically significant abnormal ECG, uncontrolled hypertension, glaucoma, symptomatic prostatic hypertrophy)
* Cancer that has not been in complete remission for at least 5 years
* Treatment with investigational study drug or participation in another clinical trial or study within the last 30 days or 5 half lives

Other inclusion/exclusion criteria as defined in the protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2011-10-01 (Actual); Study Completion 2011-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics, Inc.
Locations (8):
- United States (8):
  - Pearl Investigative Site, Panama City, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Cherry Hill, New Jersey
  - Pearl Investigative Site, Summit, New Jersey
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Medford, Oregon
  - Pearl Investigative Site, Longview, Texas
  - Pearl Investigative Site, Richmond, Virginia

REFERENCES:
- [Derived] Kerwin EM, Spangenthal S, Kollar C, St Rose E, Reisner C. A phase IIb randomized, chronic-dosing, incomplete block, cross-over study of glycopyrronium, delivered via metered dose inhaler, compared with a placebo and an active control in patients with moderate-to-severe COPD. Respir Res. 2018 Mar 5;19(1):38. doi: 10.1186/s12931-018-0739-6. PMID 29506504
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4164&filename=PT001002-00_Protocol_Redacted_23JAN2018.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 9 US sites from May-October 2011. Entire period of study participation per subject was a maximum of 15 weeks. Planned target enrollment of 84 subjects.
Pre-assignment Details: This was a chronic dosing study (7 days), 3-period, 6-treatment, incomplete block, crossover study. Each subject received 3 of 6 possible treatments; each treatment period was separated by a washout period 7-28 days. By-treatment sequence tabulations of the data were not pre-specified.
Period: Overall Study
Arm/Group | All Subjects Randomized
Started | 103
GP MDI 36 µg BID | 49 (Glycopyrronium Metered Dose Inhaler)
GP MDI 18 µg BID | 49
GP MDI 9 µg BID | 49
GP MDI 4.6 µg BID | 45
Placebo MDI BID | 48
Atrovent HFA 34 µg BID | 48
Completed | 89
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Protocol discontinuation criteria | 8
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population includes all subjects who were randomized, received at least 1 dose of study treatment, and had both baseline and post-baseline efficacy data for that treatment.
Groups:
- ITT Population: ITT Population includes all subjects who were randomized, received at least 1 dose of study treatment, and had both baseline and post-baseline efficacy data for that treatment.
Arm/Group | ITT Population
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-12
Description: FEV1 AUC0-12 following chronic dosing (1 week), normalized.
Time Frame: Day 7 ( -1 hour, -30 min, 15 min, 30 min, 1 hour, 2 hours, 4 hours, 5.5 hours, 6.5 hours, 8 hours, 10 hours, 11.5 hours, and 12 hours)
Population: Modified Intent to Treat (MITT) Population includes subjects who completed at least 2 treatment periods, with minimally 1 pre-dose assessment on Day 7 for each of those 2 treatment periods with no protocol deviations believed to have a potential impact on efficacy results.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Groups:
- PT001 MDI 36 µg BID: PT001 MDI 36 µg BID.
- PT001 MDI 18 µg BID: PT001 MDI 18 µg BID.
- PT001 MDI 9 µg BID: PT001 MDI 9 µg BID
- PT001 MDI 4.6 µg BID: PT001 MDI 4.6 µg BID.
- Ipratropium Bromide HFA Inhalation Aerosol: Ipratropium Bromide HFA Inhalation Aerosol 34 µg QID.
- Placebo MDI BID: Placebo MDI BID.
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 40 | 41 | 41 | 39 | 42 | 40
Liter | 1.477 [1.418 to 1.537] | 1.497 [1.437 to 1.556] | 1.443 [1.385 to 1.501] | 1.514 [1.456 to 1.572] | 1.465 [1.405 to 1.524] | 1.323 [1.263 to 1.382]

2. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 1
Description: Highest value of FEV1 post-dose minus baseline on Day 1 (baseline-adjusted)
Time Frame: Day 1
Population: MITT Population includes subjects who completed at least 2 treatment periods, with minimally 1 pre-dose assessment on Day 7 for each of those 2 treatment periods with no protocol deviations believed to have a potential impact on efficacy results.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 46 | 44 | 41 | 44 | 46
Liter | 0.245 (0.0252) [0.195 to 0.295] | 0.221 (0.0247) [0.172 to 0.270] | 0.181 (0.0256) [0.130 to 0.232] | 0.204 (0.0206) [0.153 to 0.255] | 0.250 (0.0258) [0.198 to 0.301] | 0.071 (0.0251) [0.021 to 0.120]

3. Secondary Outcome: Time to Onset of Action ( ≥10% Improvement in FEV1) on Day 1
Description: Time to onset of action ( ≥10% improvement in FEV1)
Time Frame: Day 1 (15 min, 30 min, 1 hour, 2 hours)
Population: as for outcome 2
Measure: Number; unit: % of subjects
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 44 | 45 | 43 | 40 | 44 | 45
% of subjects
  15 minutes | 32 | 31 | 19 | 25 | 48 | 7
  30 minutes | 32 | 18 | 7 | 20 | 25 | 9
  1 hour | 5 | 11 | 23 | 8 | 9 | 4
  2 hours | 2 | 13 | 14 | 15 | 2 | 13
  No onset within 2 hours | 30 | 27 | 37 | 33 | 16 | 67

4. Secondary Outcome: Proportion of Subjects Achieving at Least 12% Improvement in FEV1 on Day 1
Description: Proportion of subjects achieving at least 12% improvement in FEV1 (relative to baseline)
Time Frame: Day 1
Population: MITT Population: This includes subjects who completed at least 2 treatment periods, with minimally 1 pre-dose assessment on Day 7 for each of those 2 treatment periods with no protocol deviations believed to have a potential impact on efficacy results.
Measure: Number; unit: Percent
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 46 | 44 | 41 | 45 | 46
Percent | 66.67 | 58.70 | 52.27 | 60.98 | 77.78 | 17.39

5. Secondary Outcome: Peak Change From Baseline in IC on Day 1
Description: Peak change from baseline in Inspiratory Capacity (IC) on Day 1 (mean of 1 and 2 hours post-dose minus baseline on Day 1)
Time Frame: Day 1
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 45 | 44 | 41 | 45 | 46
Liter | 0.240 (0.0379) [0.165 to 0.316] | 0.276 (0.0377) [0.201 to 0.351] | 0.185 (0.0374) [0.111 to 0.259] | 0.187 (0.0380) [0.111 to 0.262] | 0.252 (0.0396) [0.173 to 0.330] | 0.040 (0.0385) [-0.036 to 0.117]

6. Secondary Outcome: Change From Baseline in Morning Pre-dose FEV1 on Day 7
Description: Change from baseline in morning pre-dose FEV1
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 43 | 46
Liter | 0.088 (0.0246) [0.039 to 0.136] | 0.075 (0.0245) [0.027 to 0.124] | 0.010 (0.0248) [-0.039 to 0.059] | 0.084 (0.0247) [0.035 to 0.133] | -0.088 (0.0256) [-0.138 to -0.037] | -0.043 (0.0246) [-0.092 to 0.006]

7. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 7
Description: Peak change from baseline in FEV1
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 43 | 44
Liter | 0.242 (0.0303) [0.181 to 0.302] | 0.224 (0.0300) [0.164 to 0.284] | 0.223 (0.0307) [0.162 to 0.285] | 0.238 (0.0308) [0.176 to 0.300] | 0.225 (0.0307) [0.164 to 0.287] | 0.070 (0.0305) [0.009 to 0.131]

8. Secondary Outcome: Peak Change From Baseline in IC on Day 7
Description: Peak change from baseline in IC
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 45 | 45 | 43 | 41 | 43 | 44
Liters | 0.213 (0.0416) [0.130 to 0.295] | 0.189 (0.0411) [0.107 to 0.271] | 0.161 (0.0424) [0.077 to 0.245] | 0.192 (0.0426) [0.107 to 0.277] | 0.191 (0.0424) [0.106 to 0.275] | -0.029 (0.0419) [-0.112 to 0.055]

9. Secondary Outcome: Change From Baseline in 12-hour Post-dose Trough FEV1 on Day 7
Description: Change from baseline in 12-hour post-dose trough FEV1
Time Frame: Day 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo MDI BID
Number analyzed (Participants) | 40 | 41 | 41 | 39 | 42 | 41
Liters | 0.018 (0.0313) [-0.045 to 0.080] | 0.079 (0.0304) [0.018 to 0.139] | 0.004 (0.0306) [-0.057 to 0.065] | 0.077 (0.0307) [0.016 to 0.139] | -0.041 (0.0311) [-0.103 to 0.021] | -0.054 (0.0316) [-0.117 to 0.009]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent up to the follow-up phone call 7-14 days after last dose of study drug.
Description: Safety population included all participants who received at least one dose of investigational drug and had safety data available; participants were included in safety population according to the investigational drug received
Groups:
- Placebo BID: Placebo BID.
Arm/Group | PT001 MDI 36 µg BID | PT001 MDI 18 µg BID | PT001 MDI 9 µg BID | PT001 MDI 4.6 µg BID | Ipratropium Bromide HFA Inhalation Aerosol | Placebo BID
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 1/45 | 1/48 | 0/48
Other Adverse Events (participants affected / at risk) | 1/49 | 2/49 | 4/49 | 4/45 | 3/48 | 1/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PT001 MDI 36 µg BID (N=49) | PT001 MDI 18 µg BID (N=49) | PT001 MDI 9 µg BID (N=49) | PT001 MDI 4.6 µg BID (N=45) | Ipratropium Bromide HFA Inhalation Aerosol (N=48) | Placebo BID (N=48)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PT001 MDI 36 µg BID (N=49) | PT001 MDI 18 µg BID (N=49) | PT001 MDI 9 µg BID (N=49) | PT001 MDI 4.6 µg BID (N=45) | Ipratropium Bromide HFA Inhalation Aerosol (N=48) | Placebo BID (N=48)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 4 (4) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.